CLINICAL TRIAL: NCT00401115
Title: A Phase 1, Open-Label, Dose-Escalation Clinical Study to Assess the Safety and Tolerability of MS-R001 in Patients With Diabetic Macular Edema Secondary to Diabetic Retinopathy
Brief Title: Safety and Tolerability of MS-R001 in Patients With Diabetic Macular Edema Secondary to Diabetic Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Mihoko Suzuki Harr/Associate Director, Clinical Affairs, Santen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR-001
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subconjunctival injection
  Interventions: Drug: MS-R001 (rapamycin)
- 2 (Experimental): Intraocular injection
  Interventions: Drug: MS-R001 (rapamycin)

INTERVENTIONS:
Drug: MS-R001 (rapamycin) — Subconjunctival injection in various dosages
  Other Names: sirolimus
  Arms: 1
Drug: MS-R001 (rapamycin) — Intraocular injection in various dosages
  Other Names: sirolimus
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and tolerability of MS-R001 at escalating doses in patients with diabetic macular edema secondary to diabetic retinopathy

ELIGIBILITY:
Inclusion Criteria include but are not limited to:

* Diagnosed with diabetes mellitus
* Visual acuity of 20/40 to 20/200 in study eye

Exclusion Criteria include but are not limited to:

* Any other ocular disease that could compromise vision in the study eye
* Intraocular surgery of the study eye within 90 days prior to study start
* Capsulotomy of the study eye within 30 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by visual acuity, intraocular pressure, slit lamp and indirect ophthalmoscope | 12 months

SECONDARY OUTCOMES:
Visual Acuity | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Dugel, M.D., Principal Investigator — Retina Consultants of Arizona; Wayne Solley, M.D., Principal Investigator — Texas Retina Associates
Locations (2):
- United States (2):
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Texas Retina Associates, Arlington, Texas